CLINICAL TRIAL: NCT06925815
Title: Pregnancy Cohort Study: Pregnancy as a Window to Future Health
Acronym: PregWin
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 34-264 ex 21/22
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Healthy Pregnant Women; Obese Pregnant Women; Gestational Diabetes
Keywords: pregnancy; deep phenotyping; maternal metabolism; body composition; longitudinal pregnancy cohort study; fetal growth; obesity in pregnancy; neonatal adiposity; gestational weight gain; gestational diabetes; cardiovascular health
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Obesity; Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal samples: serum, ccfDNA (PAXgene), urine, saliva, vaginal swabs (at 14 wks, 24 wks and 37 wks of gestation, 8-12 wks post partum); cord blood samples: serum, ccfDNA (PAXgene); placenta and umbilical cord tissue; amniotic fluid (C-section); colostrum (48h postpartum); human milk (8-12 weeks post partum)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cohort study is to gain deep insights into how metabolic disorders such as obesity or diabetes during pregnancy affect the metabolic and cardiovascular health of mother and child in the short and long term.

It will investigate the following questions:

* How do maternal metabolic disorders affect pregnancy outcomes?
* How do maternal metabolic disorders affect fetal growth?
* How do maternal metabolic disorders affect the newborn's metabolism and body composition?
* How do maternal metabolic disorders during pregnancy affect breast milk composition?
* How do maternal metabolic disorders during pregnancy affect the metabolic health of the mother after birth? Participants in this study are pregnant women who will be asked to come to the clinics for three visits during their pregnancy, as well as for the delivery of their baby, and one time 2-3 months thereafter. At each visit, researchers will perform physical examinations (such as body composition measurements) and collect biological samples (blood, urine, saliva), clinical information, and lifestyle data. At birth, researchers will collect cord blood and breast milk as well as clinical data of the delivery and the health of the baby. Researchers will measure body fat in newborn babies and at 2-3 months of age.

DETAILED DESCRIPTION:
Pregnancy is a sensitive and determining period in life where maternal and environmental cues can influence mother and offspring health short and long term. Negative exposures in pregnancy can have long term consequences, such as higher risk for development or aggravation of obesity, metabolic and cardiovascular diseases. However, preventive measures such as life style interventions can be particularly effective (window of opportunity) and could mitigate disease trajectories.

During a healthy pregnancy, a multitude of fine-tuned physiological adaptations takes place to meet the demands of the developing fetus and prepare maternal organism for delivery and lactation. These physiological changes affect the maternal metabolism, cardiovascular system, immune system, microbiome, or endocrine system. Unfavorable or adverse maternal factors (e.g. endocrine, genetic, metabolic, lifestyle factors) may compromise these adaptations, promoting pregnancy complications such as gestational diabetes (GDM), hypertensive pregnancy diseases, fetal growth restriction, fetal overgrowth, or preterm birth. These pregnancy pathologies not only pose an immediate health risk to both mother and child, but also may negatively impact the longer-term cardiovascular, endocrine, and metabolic health of both.

Offspring exposed in utero to maternal diabetes, hypertensive diseases or maternal obesity are at higher risk of developing obesity, diabetes of cardiovascular disorders later in life. For the mother, each pregnancy loads a metabolic burden, which is aggravated by pregnancy complications, also increasing the mother's risk of developing metabolic or cardiovascular disease later in life.

Therefore, prediction and risk evaluation, early diagnosis and prognosis, safe (non-invasive) therapeutic strategies are urgently needed to provide intervention as early as possible (pre-conceptional, during pregnancy and postpartum) to avoid potential manifestations of long-term health problems. Due to the relatively short duration of pregnancy and the often increased health awareness of expectant mothers, pregnancy is an ideal phase to identify origins of disease, evaluate personalized diagnostic and predictive markers, as well as preventive strategies.

In the recent years, the concept of deep phenotyping during pregnancy has emerged as a means to tackle the current inadequate understanding on the pathobiology of pregnancy related diseases and heath trajectories.

The proposed pregnancy and birth cohort aims to meet this need providing comprehensive sets of biological samples, clinical data, physical measurements and life style information for deep phenotyping of pregnancy and early life. Special focus will be put on monitoring glucose metabolism throughout pregnancy and postpartum, since the standard care oGTT at 24 to 28 weeks merely detects an already manifest glucose intolerance without giving any information on potentially preconceptionally existing impaired glucose tolerance/pre-diabetes or predicting maternal hyperglycemia thereafter, in late pregnancy.

This study will be a monocentric, prospective cohort with the goal of recruiting 80-100 participants per year. The study will be conducted at the LKH Graz University Hospital, Department of Gynecology and Obstetrics, Outpatient Clinic. Women with child wish will be recruited at the Center for Assisted Reproductive Technologies (Center for Gynecologic Endocrinology and Reproductive Medicine, Kinderwunsch-Zentrum) or pregnant women attending their routine first trimester screening visits will be enrolled and followed throughout their pregnancy until 8-12 weeks postpartum. There will be up to 6 visits: (T0 preconceptional enrollment), T1 (10-14 weeks of gestation, first trimester screening/enrollment), T2 (24-28 weeks of gestation, time of routine care oGTT); T3 (34-37 weeks of gestation, late pregnancy control visit in preparation for delivery), T4 (delivery), T5 (8-12 weeks postpartum; follow-up after pregnancy complications). The study is designed to closely monitor glucose metabolism and requires participants to be fasting for blood sampling. Women will be offered an oGTT at each visit (at T2 standard of care), but may opt out.

The study will collect clinical markers and measurements of metabolic and hemodynamic parameters, as well as a comprehensive collection of biospecimens and metadata on lifestyle factors (nutrition, physical activity). Advanced methods such as maternal and infant air displacement plethysmography (BODPOD /PEAPOD) will provide accurate body composition measurements. Endothelial/vascular function is assessed by hemodynamic parameters, including pulse wave velocity measured with a Vicorder®.

ELIGIBILITY:
Inclusion Criteria:

* ongoing pregnancy prior to 14th gestational week, women with child wish; above 18 years of age, giving informed consent

Exclusion Criteria:

* gestational age > 14th week of gestation; below 18 years of age; fetal genetic anomalies /malformation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eligible for participation are women with child wish and women with an on-going pregnancy who are planning to give birth at the university hospital in Graz, Austria. Women will be recruited as soon as possible in their pregnancy, but not after the 14th week of gestation. They will be recruited through the outpatient clinics and, in case of women with child wish, at the center for assisted reproductive technologies at the Department of Obstetrics and Gynecology, at Medical University Graz.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2033-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Maternal adiposity | From enrolment to 8-12 weeks post partum
  Measured as fat mass and fat-free mass by air displacement plethysmography (via BODPOD) at 10-14 weeks, 20-24 weeks and 34-37 weeks of gestation and 8-12 weeks post partum.
Maternal fasting blood glucose | from enrollment to 8-12 weeks postpartum
  Fasting blood glucose as measured in mg/mL from NaF blood tubes at 10-14 weeks, 24-24 weeks, 34-37 weeks of gestation and 8-12 postpartum.
Maternal blood pressure | From enrolment to 8-12 weeks postpartum
  Blood pressure will be measured at 10-14 weeks, 24-28 weeks and 34-37 weeks of gestation and 8-12 weeks post partum.
Maternal lipid profiles - triglycerides | From enrolment to 8-12 weeks post partum
  Analysis of serum lipid profiles: triglycerides at 3 time points during pregnancy (10-14 weeks (wks); 24-28wks; 34-37wks), and 8-12 wks postpartum.
Maternal lipid profiles: phospholipids | From enrolment to 8-12 weeks post partum
  Analysis of serum lipid profiles: phospholipids at 3 time points during pregnancy (10-14wks; 24-28wks; 34-37wks), and 8-12wks postpartum.
Maternal lipid profiles: free fatty acids | From enrolment to 8-12 weeks post partum
  Analysis of serum lipid profiles: free fatty acids at 3 time points during pregnancy (10-14wks; 24-28wks; 34-37wks), and 8-12wks postpartum.
Maternal lipid profiles: total cholesterol | From enrolment to 8-12 weeks post partum
  Analysis of serum lipid profiles: total cholesterol at 3 time points during pregnancy (10-14wks; 24-28wks; 34-37wks), and 8-12wks postpartum.
Maternal lipid profiles: HDL cholesterol | From enrolment to 8-12 weeks post partum
  Analysis of serum lipid profiles: HDL cholesterol at 3 time points during pregnancy (10-14wks; 24-28wks; 34-37wks), and 8-12wks postpartum.
Maternal lipid profiles: LDL cholesterol | From enrolment to 8-12 weeks post partum
  Analysis of serum lipid profiles: LDL cholesterol at 3 time points during pregnancy (10-14wks; 24-28wks; 34-37wks), and 8-12wks postpartum.
Maternal endothelial function | From enrolment to 8-12 weeks post partum
  measured as pulse wave velocity using a Vicorder®.
Maternal cytokine profile | From enrolment to 8-12 weeks postpartum
  Serum cytokines will be analysed by multiplexing at all visits during pregnancy and postpartum.
Gestational diabetes | From enrolment to child birth; 6 months
  assessed through 75g 2h oral glucose tolerance test performed at 24-28 weeks of gestation.
Hypertensive disorders of pregnancy | From enrolment to child birth; 6 months
  gestational hypertension and preeclampsia, assessed through medical chart review.
Neonatal body composition at birth | between delivery and 48h postpartum
  Measured as fat mass and fat-free mass by air displacement plethysmography (via PEAPOD)
Neonatal C-peptide in cord blood | at birth
  Concentrations of C-peptide in cord blood
Neonatal cytokine profile | at birth
  Neonatal inflammatory cytokines will be measured in cord blood serum collected at birth using multiplexing cytokine assays.
Neonatal epigenetic profile | at birth
  Epigenomic profile of the umbilical cord blood measured by DNA methylation

SECONDARY OUTCOMES:
Human milk oligosaccharide (HMO) profile in maternal blood | From enrolment to 8-12 weeks postpartum
  HMOs will be analysed in maternal serum by high pressure liquid chromatography (HPLC) with fluorescence detection
Human milk oligosaccharide (HMO) profile in maternal urine | From enrolment to 8-12 weeks post partum
  HMOs will be analysed in maternal serum by high pressure liquid chromatography (HPLC) with fluorescence detection
Human milk oligosaccharide (HMO) profile in cord blood | at birth
  HMOs will be analysed in umbilical cord blood serum by high pressure liquid chromatography (HPLC) with fluorescence detection
Human milk oligosaccharide (HMO) profile in breast milk | from child birth to 8-12 weeks postpartum
  HMOs will be analysed in breast milk by high pressure liquid chromatography (HPLC) with fluorescence detection
Adverse pregnancy outcome | From enrolment to child birth; 6 months
  Composite measure including gestational hypertension, preeclampsia, gestational diabetes, preterm delivery, low birth weight, assessed through medical chart review

OTHER OUTCOMES:
Maternal vaginal microbiome | From enrolment to 8-12 weeks postpartum
  From the extracted DNA, 16S rRNA genes will be amplified using specific primers for bacterial and archaeal communities. The amplicons obtained will be prepared for Illumina MiSeq Sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Jantscher-Krenn, PhD, Principal Investigator — Medical University of Graz; Herbert Fluhr, Univ.-Prof. Dr. med., Study Director — Medical University of Graz
Locations (1):
- Department of Obstetrics and Gynecology, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying results in a publication will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available starting 1 year after publication with no end date.
Access Criteria: Data access will be provided to external researchers who submit a methodologically sound proposal for secondary data analysis that is approved by the study investigators and should be submitted to the study PI.